CLINICAL TRIAL: NCT06036511
Title: Connectivity Changes Associated With Ketamine Assisted Psychotherapy for PTSD
Acronym: CONCHKAP
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per PI, this trial will not be started at UNM due to change in institutional responsibilities of the PI
Sponsor: University of New Mexico (Other)
Collaborators: The Mind Research Network (Other)
Responsible Party: Principal Investigator, Snehal Bhatt, MD, Chief, Addiction Psychiatry, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-116
Record Dates: First submitted 2023-08-03; First posted 2023-09-14 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: PTSD
Keywords: PTSD; Ketamine Assisted Psychotherapy; Brain network connectivity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: This is a single arm, open-label, prospective cohort clinical trial.
  No blinding is required for this trial.
  A total of 14 adult patients with PTSD will be recruited from UNM outpatient clinics and undergo rsfMRI and behavioral assessment prior to ketamine treatment. They will complete baseline scan at day one, a preparatory session (initial part of KAP), IM ketamine treatment, then within 24 hours, an integration session to take advantage of neuroplasticity for optimal therapeutic progress. Each participant will have two complete KAP sessions (preparation, treatment, and integration) followed by rsfMRI within approximately 24 hours, and again approximately two weeks after the completion of the second KAP session. Patients will also have repeat clinical assessments after each treatment. Changes in PTSD symptoms will be correlated with changes in connectivity at each rsfMRI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ketamine Assisted Psychotherapy [KAP] (Experimental): A total of 14 adult patients with PTSD will be recruited from UNM outpatient clinics and undergo rsfMRI and behavioral assessment prior to ketamine treatment. They will complete baseline scan at day one, a preparatory session (initial part of KAP), IM ketamine treatment, then within 24 hours, an integration session to take advantage of neuroplasticity for optimal therapeutic progress. Each participant will have two complete KAP sessions (preparation, treatment, and integration) followed by rsfMRI within approximately 24 hours, and again approximately two weeks after the completion of the second KAP session. Patients will also have repeat clinical assessments after each treatment. Changes in PTSD symptoms will be correlated with changes in connectivity at each rsfMRI.
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — This is a single arm, open-label, prospective cohort clinical trial.
  No blinding is required for this trial.
  A total of 14 adult patients with PTSD will be recruited from UNM outpatient clinics and undergo rsfMRI and behavioral assessment prior to ketamine treatment. They will complete baseline scan at day one, a preparatory session (initial part of KAP), IM ketamine treatment, then within 24 hours, an integration session to take advantage of neuroplasticity for optimal therapeutic progress. Each participant will have two complete KAP sessions (preparation, treatment, and integration) followed by rsfMRI within approximately 24 hours, and again approximately two weeks after the completion of the second KAP session. Patients will also have repeat clinical assessments after each treatment. Changes in PTSD symptoms will be correlated with changes in connectivity at each rsfMRI.
  Other Names: KAP

SUMMARY:
The goal of this clinical trial is to learn about the effects of Ketamine Assisted Psychotherapy [KAP] on individuals with Post Traumatic Stress Disorder [PTSD]. The main questions it aims to answer are:

1. Does KAP improve symptoms of PTSD?
2. What changes in brain network connectivity are seen with KAP?

DETAILED DESCRIPTION:
A total of 14 adult patients with PTSD will be recruited from UNM outpatient clinics and undergo rsfMRI and behavioral assessment prior to ketamine treatment. They will complete baseline scan at day one, a preparatory session (initial part of KAP), IM ketamine treatment, then within 24 hours, an integration session to take advantage of neuroplasticity for optimal therapeutic progress. Each participant will have two complete KAP sessions (preparation, treatment, and integration) followed by rsfMRI within approximately 24 hours, and again approximately two weeks after the completion of the second KAP session. Patients will also have repeat clinical assessments after each treatment. Changes in PTSD symptoms will be correlated with changes in connectivity at each rsfMRI.

ELIGIBILITY:
Inclusion Criteria:

* Participants may be eligible for enrollment if all the following inclusion criteria apply within the thirty days prior to first ketamine administration session:

Between the ages of 18 to 65 years old.

Meet DSM-5 criteria for Port-Traumatic Stress Disorder [PTSD] based on clinical interview.

Able to provide informed consent.

Are proficient in reading and speaking English.

Agree to refrain from using stimulants during the day of the medication session.

Agree to refrain from alcohol and cannabis for 24 hours before and the day of medication session.

Subjects taking other psychotropic medications (e.g. anti-depressants, anxiolytics, methadone, buprenorphine, naltrexone) must be maintained on a stable dose for at least four weeks before study initiation.

Agree to not operate a car or any other heavy equipment for the rest of the day after the ketamine administration.

If necessary, are willing to be contacted via telephone on a daily basis by the therapist or team after each experiential session.

Able to identify one or two caregiver support persons who can drive participant home, stay with them overnight, be reached by the team, and provide collateral information as needed.

Willing to inform the investigator within 48 hours if any medical conditions occur or procedures are planned.

Exclusion Criteria:

* Participants will be excluded from the study if any of the following criteria apply:

They are considered an immediate suicide risk by clinician assessment or felt to be likely to require hospitalization during the study.

Have had a psychiatric or medical hospitalization, or an Emergency Department visit, within four weeks of the study entry.

Subjects who meet DSM-5 criteria for current bipolar disorder based on clinical interview.

Subjects who meet DSM-5 criteria for current or history of psychotic spectrum disorders based on clinical interview.

Subjects meeting DSM-5 criteria for current substance use disorder (i.e., not in early or sustained remission) other than tobacco use disorder.

Subjects who report use of ketamine >20 times in the past or who meet DSM-5 criteria for Other Hallucinogen Use Disorder due to ketamine use including subjects who are currently in early or sustained remission.

Women who are pregnant or nursing, and women who do not consent to use methods of highly effective birth control during the study.

Subjects with hypertension as defined by a baseline visit systolic blood pressure (SBP) >140 mmHg or a diastolic blood pressure (DBP) >90 mmHg.

A history of allergic or other adverse reaction to ketamine (or its excipients).

Clinically significant physical exam findings or self-reported medical conditions for which a transient increase in blood pressure could be significantly detrimental (e.g. glaucoma, aneurysmal disease, cardiovascular disease, or end-stage renal disease).

QTc will be measured in all subjects and those with QTc 450ms or longer will be excluded.

High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, antisocial behavior, serious current stressors, lack of meaningful social support).

Documented evidence of significant renal or hepatic dysfunction at screening. Significantly impaired liver function is defined as 1) Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 5 × upper limit of normal (ULN); 2) ALT or AST > 3 × ULN with concomitant total bilirubin > 2.0 × ULN; or 3) ALT or AST ≥ 3 × ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia.

Blood pressure will be monitored at all subsequent visits, and participants will receive study medication only if blood pressure is less than or equal to 140 systolic, 90 diastolic at safety screening on the day of the drug administration sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical outcome: PTSD severity | 14-21 days
  as defined by change in score on Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) following KAP treatments (Assessment Visit 3) compared to baseline (Assessment Visit 1).
Imaging Outcome: Changes in functional connectivity | 28-35 days
  change in the functional connectivity between vmPFC and amygdala from Baseline to Assessment Visit 4 as measured by fMRI.

SECONDARY OUTCOMES:
Depression severity | 14-21 days
  Improvement in depression, as indicated by reduced Montgomery-Asberg Depression Rating Scale (MADRS), following KAP treatments (Assessment Visit 3) compared to baseline (Assessment Visit 1).
Persisting PTSD effect | 28-35 days
  The changes in score on Clinician-Administered PTSD Scale for DSM-5 (CAPS-5).
Correlation of clinical and imaging outcomes | 28-35 days
  Change in connectivity between the vmPFC and amygdala from Assessment Visit 1 to Assessment Visit 4 with degree of PTSD symptom change.
Persisting MDD effect | 28-35 days
  Concurrent MDD (MADRS) will persist at last evaluation two weeks after completion of active treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Bhatt, MD, Principal Investigator — UNM
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drozdz SJ, Goel A, McGarr MW, Katz J, Ritvo P, Mattina GF, Bhat V, Diep C, Ladha KS. Ketamine Assisted Psychotherapy: A Systematic Narrative Review of the Literature. J Pain Res. 2022 Jun 15;15:1691-1706. doi: 10.2147/JPR.S360733. eCollection 2022. PMID 35734507
- [Background] Joneborg I, Lee Y, Di Vincenzo JD, Ceban F, Meshkat S, Lui LMW, Fancy F, Rosenblat JD, McIntyre RS. Active mechanisms of ketamine-assisted psychotherapy: A systematic review. J Affect Disord. 2022 Oct 15;315:105-112. doi: 10.1016/j.jad.2022.07.030. Epub 2022 Jul 26. PMID 35905796
- [Background] Dore J, Turnipseed B, Dwyer S, Turnipseed A, Andries J, Ascani G, Monnette C, Huidekoper A, Strauss N, Wolfson P. Ketamine Assisted Psychotherapy (KAP): Patient Demographics, Clinical Data and Outcomes in Three Large Practices Administering Ketamine with Psychotherapy. J Psychoactive Drugs. 2019 Apr-Jun;51(2):189-198. doi: 10.1080/02791072.2019.1587556. Epub 2019 Mar 27. PMID 30917760
- [Background] Feder A, Costi S, Rutter SB, Collins AB, Govindarajulu U, Jha MK, Horn SR, Kautz M, Corniquel M, Collins KA, Bevilacqua L, Glasgow AM, Brallier J, Pietrzak RH, Murrough JW, Charney DS. A Randomized Controlled Trial of Repeated Ketamine Administration for Chronic Posttraumatic Stress Disorder. Am J Psychiatry. 2021 Feb 1;178(2):193-202. doi: 10.1176/appi.ajp.2020.20050596. Epub 2021 Jan 5. PMID 33397139
- [Background] Ionescu DF, Felicione JM, Gosai A, Cusin C, Shin P, Shapero BG, Deckersbach T. Ketamine-Associated Brain Changes: A Review of the Neuroimaging Literature. Harv Rev Psychiatry. 2018 Nov/Dec;26(6):320-339. doi: 10.1097/HRP.0000000000000179. PMID 29465479
- [Background] Norbury A, Rutter SB, Collins AB, Costi S, Jha MK, Horn SR, Kautz M, Corniquel M, Collins KA, Glasgow AM, Brallier J, Shin LM, Charney DS, Murrough JW, Feder A. Neuroimaging correlates and predictors of response to repeated-dose intravenous ketamine in PTSD: preliminary evidence. Neuropsychopharmacology. 2021 Dec;46(13):2266-2277. doi: 10.1038/s41386-021-01104-4. Epub 2021 Jul 31. PMID 34333555
- [Background] Krystal JH, Abdallah CG, Averill LA, Kelmendi B, Harpaz-Rotem I, Sanacora G, Southwick SM, Duman RS. Synaptic Loss and the Pathophysiology of PTSD: Implications for Ketamine as a Prototype Novel Therapeutic. Curr Psychiatry Rep. 2017 Aug 26;19(10):74. doi: 10.1007/s11920-017-0829-z. PMID 28844076
- [Background] Patel R, Spreng RN, Shin LM, Girard TA. Neurocircuitry models of posttraumatic stress disorder and beyond: a meta-analysis of functional neuroimaging studies. Neurosci Biobehav Rev. 2012 Oct;36(9):2130-42. doi: 10.1016/j.neubiorev.2012.06.003. Epub 2012 Jul 2. PMID 22766141
- [Background] Sheynin J, Liberzon I. Circuit dysregulation and circuit-based treatments in posttraumatic stress disorder. Neurosci Lett. 2017 May 10;649:133-138. doi: 10.1016/j.neulet.2016.11.014. Epub 2016 Nov 12. PMID 27845239
- [Background] Stopyra MA, Simon JJ, Rheude C, Nikendei C. Pathophysiological aspects of complex PTSD - a neurobiological account in comparison to classic posttraumatic stress disorder and borderline personality disorder. Rev Neurosci. 2022 Aug 8;34(1):103-128. doi: 10.1515/revneuro-2022-0014. Print 2023 Jan 27. PMID 35938987
- [Background] Fonzo GA, Goodkind MS, Oathes DJ, Zaiko YV, Harvey M, Peng KK, Weiss ME, Thompson AL, Zack SE, Lindley SE, Arnow BA, Jo B, Rothbaum BO, Etkin A. Amygdala and Insula Connectivity Changes Following Psychotherapy for Posttraumatic Stress Disorder: A Randomized Clinical Trial. Biol Psychiatry. 2021 May 1;89(9):857-867. doi: 10.1016/j.biopsych.2020.11.021. Epub 2020 Dec 8. PMID 33516458